CLINICAL TRIAL: NCT05349331
Title: Watch and Wait and Surgical Treatment for Clinical Complete Responders After Non-Curative Therapy for Hepatocellular Carcinoma: A Phase II Randomized Clinical Trial
Brief Title: Watch and Wait and Surgical Treatment for Clinical Complete Responders After Non-Curative Therapy for Hepatocellular Carcinoma
Acronym: WATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Binkui Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-119-X01
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Conversion Reaction
MeSH Terms: conditions — Carcinoma, Hepatocellular; Conversion Disorder | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection group (Experimental): Surgical resection group: The patients underwent liver cancer resection and were followed up regularly after surgery.
  Interventions: Procedure: Liver Resection
- Non-surgical resection group (No Intervention): Stop hepatic artery interventional therapy (chemoembolization/infusion chemotherapy), continue the original targeted and immunotherapy for no more than 1 year

INTERVENTIONS:
Procedure: Liver Resection — Surgical resection treatment: laparoscopic or open liver resection is performed, and targeted and immunotherapy are not continued after surgery.
  Arms: Resection group

SUMMARY:
Hepatocellular carcinoma (HCC) accounts for more than 90% of primary liver cancers and is the sixth most common cancer in the world and ranked third in mortality. Most patients with HCC are diagnosed at an advanced stage and miss the opportunity for radical surgical resection, therefore, most patients receive mainly non-curative local and systemic treatments.

Anti-angiogenic drugs with immunotherapy for unresectable HCC has achieved an objective response rate of about 30%. In addition, transarterial hepatic artery chemoembolization and hepatic artery infusion chemotherapy have further increased the objective response rate and depth of tumor regression. For patients with initially unresectable HCC, conversion therapy can result tumor shrinkage and downstaging, ultimately allowing patients the opportunity to undergo resection. However, it raise the question of whether surgical resection of the tumor is still necessary after achieving clinical complete response? On the one hand, some researchers believe that as long as resection is feasible, the tumor must be completely removed. Viable tumor cells may still remain and become a source of tumor recurrence. On the other hand, some researchers believe that patients who achieve clinical complete response after conversion therapy can consider a non-surgical watch and wait strategy. Whether the inactive lesions with clinical complete response still require surgical resection is still inconclusive. This study compared the efficacy and safety of surgical resection versus non-surgical resection in the treatment of hepatocellular carcinoma patients who achieved clinical complete response after hepatic arterial intervention (chemoembolization/infusion chemotherapy) combined with targeted and immunosuppressive therapy. It is expected to provide reliable clinical evidence support for guiding the treatment of such patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Patients with clinical diagnosis of hepatocellular carcinoma without extrahepatic metastasis, and two liver surgeons evaluated as unresectable.
* AFP≥400ug/L or PIVKA-II≥1000mAU/mL before initial treatment.
* Initial treatment is hepatic arterial intervention (chemoembolization/infusion chemotherapy), combined targeted therapy (sorafenib, lenvatinib, donafenib, apatinib, bevacizumab) and immune checkpoint inhibitor therapy (PD-1\PD-L1).
* After transarterial infusion chemotherapy combined with targeted and immunotherapy treatment, the tumor evaluation is clinical complete response, that is, the following two criteria are met: 1. Two consecutive imaging assessments (one month apart) tumor complete response (CR, mRECIST) standard) 2. Two consecutive tumor markers (one month apart) AFP and PIVKA-II ≤ the upper limit of the normal value
* The patients with clinical complete response were evaluated by two liver surgeons as resectable.
* Normal hematological function (platelets>75×109/L; leukocytes>3.0×109/L; neutrophils>1.5×109/L)
* Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), transaminases ≤ 3 times ULN
* No ascites, normal coagulation function, albumin≥30g/L
* Child-Pugh class A
* Serum creatinine less than 1.5 times the upper limit of normal (ULN)
* ECOG score 0-1
* Life expectancy > 3 months

Exclusion Criteria:

* Received other tumor treatments other than hepatic artery interventional therapy, targeted and immunotherapy
* Any of the following conditions within the first 12 months of the study: myocardial infarction, severe/unstable angina, coronary artery bypass grafting, congestive heart failure, cerebrovascular accident (including transient ischemic attack), Pulmonary embolism; ongoing: arrhythmia of grade ≥2 by NCI-CTCAE criteria, QTc prolongation (>450 ms in men, >470 ms in women);
* Renal insufficiency requires peritoneal dialysis or hemodialysis;
* Serious dysfunction of other important organs;
* A second primary malignant tumor was diagnosed in the past;
* Known or new evidence of brain or leptomeningeal lesions; Hemophilia or bleeding tendency, taking anticoagulation therapy such as coumarin derivatives in therapeutic doses;
* Pregnant or lactating women, all female patients of childbearing potential must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative;
* History of previous organ transplantation;
* Known HIV infection;
* Allergy to chemotherapy drugs;
* Patients with other serious acute or chronic physical or psychiatric diseases or abnormal laboratory tests that may increase the risk associated with participating in the study, or may interfere with the interpretation of the study results or the investigators consider unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 24 months
  Resection group: time from start of randomization to first recurrence/death. Non-resection group: time from start of randomization to first tumor progression/death.

SECONDARY OUTCOMES:
Time to treatment failure | 24 months
  Defined as the time from randomization to the first documented treatment failure (ie, local recurrence or progression or death from any cause).
Overall survival | 24 months
  defined as the time from randomization to death from any cause.
pCR rate in surgery group | 24 months
  Pathological complete response (pCR) was defined as the absence of residual viable tumor cells on hematoxylin and eosin staining on completely resected tumor specimen sections.

OTHER OUTCOMES:
Correlation of serum tumor molecular marker with survival | 24 months
  Correlation of serum tumor molecular marker methylation level with pCR in surgery group and tumor progression in non-surgery group.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China